CLINICAL TRIAL: NCT04383704
Title: Effect of MIND Diet Intervention on Cognitive Performance and Brain Structure in Healthy Obese Women: A Randomized Controlled Trial
Brief Title: MIND Diet Intervention and Cognitive Performance
Acronym: MIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammad Hassan Eftekhari, PHD. professor of clinical nutrition (clinical nutrition, school of nutrition and food science), Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IR.SUMS.REC.1397.759
Record Dates: First submitted 2020-05-05; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- calorie-restricted modified MIND diet (Experimental): This arm received instruction in modifying the content of their diet to meet MIND pattern guidelines.
  Interventions: Other: New Dietary pattern ( Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND))
- calorie-restricted standard control diet (Active Comparator): They instructed to calorie-restricted diet alone.
  Interventions: Other: New Dietary pattern ( Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND))

INTERVENTIONS:
Other: New Dietary pattern ( Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND)) — A new brain-protection pattern that has been designed after the Mediterranean and DASH diet to improve some of their dietary factors to have the highest impact on brain health and cognitive performance.

SUMMARY:
This single-center, randomized trial examined the effect of MIND diet intervention on cognition and brain structure changes of healthy obese women over three months. The intervention group was lea to calorie-restricted modified by the MIND diet, and the control group received a calorie-restricted standard diet. The primary end-point was an assessment of cognitive performances measured with a comprehensive cognitive test battery. Secondary end-points were voxel-based morphometry to quantify the differences in brain structures. Our results revealed MIND diet could improve working memory, verbal recognition memory, and attention, more in comparison with the control group. Results also suggest that an increase in inferior frontal gyrus in the MIND diet group. Our study, for the first time, underlined that good adherence to the MIND diet as well as calorie restriction could reverse the destructive effect of obesity on cognition.

ELIGIBILITY:
Inclusion Criteria:

* Middle-aged women (40-60 years),
* Without any metabolic complication,
* BMI 30-35 kg/m2,
* MMSE ≥ 24,
* And no history of severe untreated medical, neurological, and psychiatric diseases which may interfere with the study intervention.

Exclusion Criteria:

* Have gastrointestinal problems,
* Participate in weight loss programs,
* Use weight loss drugs in the last three months,
* Had not wholly followed the dietary pattern,
* Became pregnant,
* And undergo special medical treatments during a three months study.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Assessment of changes in cognitive performance tests measured by a complex paper cognitive battery at the baseline and after three months follow up. | Baseline and after three months.
  All of the participants were tested on a complex paper-based battery of neurocognitive tests to examine changes in cognitive performance in different domains at baseline and after three months follow up. These tests include Forward Digit Span Task (FDST), Backward Digit Span Task (BDST), Letter Number Sequencing Task (LNST), Symbol Digit Modality Task (SDMT), Auditory Verbal Learning Test (AVLT) and Stroop task.

SECONDARY OUTCOMES:
Assessment of changes in brain structures measured by Magnetic Resonance Imaging (MRI) baseline and after three months follow up. | Baseline and after three months.
  Magnetic Resonance Imaging (MRI) was carried out to quantify the differences in brain structure changes baseline, and after three months follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Shiraz University of Medical Science, Shiraz, Fars, Iran

REFERENCES:
- [Derived] Arjmand G, Abbas-Zadeh M, Eftekhari MH. Effect of MIND diet intervention on cognitive performance and brain structure in healthy obese women: a randomized controlled trial. Sci Rep. 2022 Feb 21;12(1):2871. doi: 10.1038/s41598-021-04258-9. PMID 35190536